CLINICAL TRIAL: NCT00565266
Title: Asthma Clinical Research Network (ACRN) Trial - Tiotropium Bromide as an Alternative to Increased Inhaled Corticosteroid in Patients Inadequately Controlled on a Lower Dose of Inhaled Corticosteroid (TALC)
Acronym: TALC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 547; U10HL074206 (NIH); U10HL074208 (NIH); U10HL074073 (NIH); U10HL074227 (NIH); U10HL074225 (NIH); U10HL074204 (NIH); U10HL074218 (NIH); U10HL074212 (NIH); U10HL074231 (NIH)
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Tio + 1xICS || LABA + 1xICS || 2xICS (Experimental): Participants will take part in three 16-week treatment periods, which will occur in the following order:
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
  Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive beclomethasone dipropionate 80 mcg twice daily (1xICS).
  Interventions: Drug: tiotropium bromide; Drug: salmeterol xinafoate; Drug: beclomethasone dipropionate
- TIO + 1xICS || 2xICS || LABA + 1xICS (Experimental): Participants will take part in three 16-week treatment periods, which will occur in the following order:
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive beclomethasone dipropionate 80 mcg twice daily (1xICS).
  Interventions: Drug: tiotropium bromide; Drug: salmeterol xinafoate; Drug: beclomethasone dipropionate
- LABA + 1xICS || Tio + 1xICS || 2xICS (Experimental): Participants will take part in three 16-week treatment periods, which will occur in the following order:
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
  Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive beclomethasone dipropionate 80 mcg twice daily (1xICS).
  Interventions: Drug: tiotropium bromide; Drug: salmeterol xinafoate; Drug: beclomethasone dipropionate
- LABA + 1xICS || 2xICS || Tio + 1xICS (Experimental): Participants will take part in three 16-week treatment periods, which will occur in the following order:
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive beclomethasone dipropionate 80 mcg twice daily (1xICS).
  Interventions: Drug: tiotropium bromide; Drug: salmeterol xinafoate; Drug: beclomethasone dipropionate
- 2xICS || Tio + 1xICS| || LABA + 1xICS (Experimental): Participants will take part in three 16-week treatment periods, which will occur in the following order:
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive beclomethasone dipropionate 80 mcg twice daily (1xICS).
  Interventions: Drug: tiotropium bromide; Drug: salmeterol xinafoate; Drug: beclomethasone dipropionate
- 2xICS || LABA + 1xICS || Tio + 1xICS (Experimental): Participants will take part in three 16-week treatment periods, which will occur in the following order:
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive beclomethasone dipropionate 80 mcg twice daily (1xICS).
  Interventions: Drug: tiotropium bromide; Drug: salmeterol xinafoate; Drug: beclomethasone dipropionate

INTERVENTIONS:
Drug: tiotropium bromide — tiotropium bromide inhalation powder 18 mcg once daily
  Other Names: SPIRIVA® HandiHaler®
Drug: salmeterol xinafoate — salmeterol xinafoate inhalation powder 50 mcg twice daily
  Other Names: Serevent® Diskus®
Drug: beclomethasone dipropionate — beclomethasone dipropionate 80 mcg twice daily (1xICS) or 160 mcg twice daily (2xICS)
  Other Names: QVAR® Inhalation Aerosol

SUMMARY:
Typically, people with asthma are initially prescribed a low dose of inhaled corticosteroid (ICS) medication to control asthma symptoms. If a low dose of ICS is ineffective at controlling symptoms, the addition of a second controller medication is recommended. This study will examine the effectiveness of the medication tiotropium bromide combined with a low dose of ICS at maintaining asthma control in people with moderately severe asthma.

DETAILED DESCRIPTION:
National and international asthma treatment guidelines recommend ICS as the initial controller therapy for people with asthma who are in need of daily treatment with a controller medication. If treatment with low to moderate doses of ICS is not sufficient to gain and maintain asthma control, current guidelines recommend adding a second controller medication rather than increasing the dose of ICS. Current options for the second medication include a long-acting beta-agonist, a leukotriene modifier, or theophylline. It is possible that other medications, not yet tested, could fill the role of the second controller medication. Tiotropium bromide is a medication that is used to treat chronic obstructive pulmonary disease (COPD). It works by relaxing and opening the air passages to the lungs to make breathing easier. For people with asthma, the addition of tiotropium bromide may be a good option as a second controller medication. The purpose of this study is to determine if combining tiotropium bromide with a low dose of ICS is more effective than doubling the dose of ICS in people with moderately severe asthma. This study will also examine whether the addition of tiotropium bromide to low dose ICS is as effective as the addition of a long-acting beta-agonist at maintaining asthma control.

This study will begin with a 4-week run-in period during which participants will be monitored while they use an inhaler containing a low dose of ICS medication. Next, participants will be assigned to take part in either the TALC study or the Best Adjustment Strategy for Asthma in Long Term (BASALT) study, which is a separate Asthma Clinical Research Network (ACRN) study.

All TALC participants will then undergo three 16-week treatment periods, which will include the following:

* tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
* salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
* beclomethasone dipropionate 160 mcg twice daily (2xICS)

The order in which the three treatment periods will occur will be randomly assigned for each participant. Each of the three 16-week treatment periods will consist of 14 weeks of treatment followed by a 2-week washout period, in which participants will receive a single does of ICS. Study visits will occur at baseline and Weeks 2 and 4 of the 4-week run-in period, and at Weeks 4, 9, 14, and 16 of each 16-week treatment period. Spirometry tests to measure lung function will occur at each study visit and exhaled nitric oxide testing and questionnaires to assess asthma control and symptoms will occur at most visits. During study visits at Week 4 of the run-in period and Week 14 of each treatment period, lung function measurements, sputum collection, questionnaires to assess asthma quality-of-life, and measurements of sleep and daytime alertness will all occur. Participants will also record asthma symptoms, peak flow measurements, and medication usage in a daily diary.

ELIGIBILITY:
Inclusion Criteria for TALC and BASALT Studies:

* Clinical history consistent with asthma
* Forced expiratory volume in one second (FEV1) greater than 40% of predicted value
* Asthma confirmed by one of the following two criteria:

  1. Beta-agonist reversibility to 4 puffs albuterol of at least 12% OR
  2. Methacholine provocative concentration at 20% (PC20) of 8 milligrams per milliliter (mg/mL) or less when not on an inhaled corticosteroid (ICS), or 16 mg/mL or less when on an ICS
* Need for daily controller therapy (i.e., ICS, leukotriene modifiers, and/or long-acting beta-agonists) based on one or more of the following criteria:

  1. Received prescription for or used asthma controller within the 12 months prior to study entry OR
  2. Experienced symptoms for more than twice a week and not on asthma controller
* If on inhaled steroids (any drug at any dose not exceeding the equivalent of 1000 micrograms (mcg) of fluticasone daily), participant must have been on a stable dose for at least 2 weeks prior to study entry
* Non-smoker (i.e., total lifetime smoking history less than 10 pack-years; no smoking for at least 1 year prior to study entry)
* Willing to use an effective form of birth control throughout the study

Inclusion Criteria for TALC Study:

* Ability to measure morning (AM) peak expiratory flow (PEF) on schedule using electronic peak flow meter (EPFM) and to complete the study diary correctly at least 75% of the time during the interval between Weeks 2 and 4 of the run-in period
* Adherence with study medication dosing at least 75% of the time during the interval between Weeks 2 and 4 of the run-in period
* No asthma exacerbation requiring use of oral corticosteroids or additional asthma medications (including an increased dose of ICS) during the run-in period
* FEV1 greater than 40% of the predicted value

Exclusion Criteria for BASALT and TALC Studies:

* Lung disease other than asthma, including chronic obstructive pulmonary disease (COPD) and chronic bronchitis
* Established or suspected diagnosis of vocal cord dysfunction
* Significant medical illness other than asthma
* History of respiratory tract infection within the 4 weeks prior to study entry
* History of a significant asthma exacerbation within the 4 weeks prior to study entry
* History of life-threatening asthma requiring treatment with intubation and mechanical ventilation in the 5 years prior to study entry
* Hyposensitization therapy other than an established maintenance regimen
* Inability to coordinate use of the delivery devices used in the study, based on the opinion of the investigator or clinical coordinator
* Pregnant

Exclusion Criteria for TALC Study:

* Inability to coordinate use of the medication delivery devices used in the study, based on the opinion of the investigator or clinical coordinator
* Presence at Week 4 of the run-in period of any of the exclusion criteria stipulated for Week 0 of the run-in period (Note: Respiratory tract infections that do not cause the participant to meet exacerbation criteria are not considered exclusionary.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Homer A. Boushey, MD, Principal Investigator — University of California, San Francisco; Richard J. Martin, MD, Principal Investigator — National Jewish Health; Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital; Stephen I. Wasserman, MD, Principal Investigator — University of California, San Diego; Mario Castro, MD, Principal Investigator — Washington University School of Medicine; Emily A. DiMango, MD, Principal Investigator — Columbia University; Stephen P. Peters, MD, PhD, Principal Investigator — Wake Forest University Health Sciences; Monica Kraft, MD, Principal Investigator — Duke University; William J. Calhoun, MD, Principal Investigator — University of Texas; Robert F. Lemanske, MD, Principal Investigator — University of Wisconsin, Madison; Reuben M. Cherniack, MD, Study Chair — National Jewish Health
Locations (10):
- United States (10):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St. Louis, St Louis, Missouri
  - Columbia University Health Sciences, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin

REFERENCES:
- [Result] Peters SP, Kunselman SJ, Icitovic N, Moore WC, Pascual R, Ameredes BT, Boushey HA, Calhoun WJ, Castro M, Cherniack RM, Craig T, Denlinger L, Engle LL, DiMango EA, Fahy JV, Israel E, Jarjour N, Kazani SD, Kraft M, Lazarus SC, Lemanske RF Jr, Lugogo N, Martin RJ, Meyers DA, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Chinchilli VM, Bleecker ER; National Heart, Lung, and Blood Institute Asthma Clinical Research Network. Tiotropium bromide step-up therapy for adults with uncontrolled asthma. N Engl J Med. 2010 Oct 28;363(18):1715-26. doi: 10.1056/NEJMoa1008770. Epub 2010 Sep 19. PMID 20979471
- [Derived] Oba Y, Anwer S, Patel T, Maduke T, Dias S. Addition of long-acting beta2 agonists or long-acting muscarinic antagonists versus doubling the dose of inhaled corticosteroids (ICS) in adolescents and adults with uncontrolled asthma with medium dose ICS: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Aug 21;8(8):CD013797. doi: 10.1002/14651858.CD013797.pub2. PMID 37602534
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Lugogo N, Green CL, Agada N, Zhang S, Meghdadpour S, Zhou R, Yang S, Anstrom KJ, Israel E, Martin R, Lemanske RF Jr, Boushey H, Lazarus SC, Wasserman SI, Castro M, Calhoun W, Peters SP, DiMango E, Chinchilli V, Kunselman S, King TS, Icitovic N, Kraft M. Obesity's effect on asthma extends to diagnostic criteria. J Allergy Clin Immunol. 2018 Mar;141(3):1096-1104. doi: 10.1016/j.jaci.2017.04.047. Epub 2017 Jun 15. PMID 28624608
- [Derived] Peters SP, Bleecker ER, Kunselman SJ, Icitovic N, Moore WC, Pascual R, Ameredes BT, Boushey HA, Calhoun WJ, Castro M, Cherniack RM, Craig T, Denlinger LC, Engle LL, Dimango EA, Israel E, Kraft M, Lazarus SC, Lemanske RF Jr, Lugogo N, Martin RJ, Meyers DA, Ramsdell J, Sorkness CA, Sutherland ER, Wasserman SI, Walter MJ, Wechsler ME, Chinchilli VM, Szefler SJ; National Heart, Lung, and Blood Institute's Asthma Clinical Research Network. Predictors of response to tiotropium versus salmeterol in asthmatic adults. J Allergy Clin Immunol. 2013 Nov;132(5):1068-1074.e1. doi: 10.1016/j.jaci.2013.08.003. Epub 2013 Sep 29. PMID 24084072
- [Derived] Sutherland ER, Goleva E, Jackson LP, Stevens AD, Leung DY. Vitamin D levels, lung function, and steroid response in adult asthma. Am J Respir Crit Care Med. 2010 Apr 1;181(7):699-704. doi: 10.1164/rccm.200911-1710OC. Epub 2010 Jan 14. PMID 20075384
- See also: Click here for the Asthma Clinical Research Network Web site — http://www.arcn.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants randomized into the six-sequence crossover study. All TALC participants underwent three 16-week treatment periods:
  * tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
  * beclomethasone dipropionate 160 mcg twice daily (2xICS)
Period: Overall Study
Arm/Group | All Participants
Started | 210
Completed | 174
Not Completed | 36

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized into the six-sequence crossover study
Arm/Group | All Participants
Number analyzed (Participants) | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 207
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 69
Region of Enrollment [Number; unit: participants]
  United States | 210

OUTCOME MEASURES:

1. Primary Outcome: Change Between Week 14 and Week 0 in the Morning (AM) Peak Expiratory Flow (PEF)
Time Frame: AM PEF was measured daily during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Groups:
- Tio + 1xICS: tiotropium bromide inhalation powder 18 mcg once daily (Tio) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
- LABA + 1xICS: salmeterol xinafoate inhalation powder 50 mcg twice daily (LABA) plus beclomethasone dipropionate 80 mcg twice daily (1xICS)
- 2xICS: beclomethasone dipropionate 160 mcg twice daily (2xICS)
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
Liters per minute | 24.4 (4.2) | 18.0 (3.2) | -1.4 (3.5)

2. Secondary Outcome: Change Between Week 14 and Week 0 in the Forced Expiratory Volume in One Second (FEV1)
Time Frame: FEV1 was measured on four occasions during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
liters | 0.12 (0.025) | 0.01 (0.025) | 0.02 (0.025)

3. Secondary Outcome: Change Between Week 14 and Week 0 in Asthma Symptoms
Description: Asthma symptoms were recorded as 0 (absent = no symptom )
  1. (mild = symptom was minimally troublesome, i.e. not sufficient to interfere with normal daily activity or sleep)
  2. (moderate = symptom was sufficiently troublesome to interfere with normal daily activity or sleep)
  3. (severe = symptom was so severe as to prevent normal activity and/or sleep )
Time Frame: Asthma symptoms were measured daily during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
units on a scale | -0.09 (0.018) | -0.04 (0.018) | 0.03 (0.018)

4. Secondary Outcome: Change Between Week 14 and Week 0 in the Asthma Quality-of-life Questionnaire Score
Description: Scores on the Asthma Quality-of-Life Questionnaire range from 1 to 7, with a higher score indicating a better quality of life.
Time Frame: The asthma quality-of-life questionnaire score was measured on four occasions during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
units on a scale | 0.15 (0.058) | 0.28 (0.050) | 0.05 (0.052)

5. Secondary Outcome: Change Between Week 14 and Week 0 in the Asthma Control Questionnaire Score
Description: Scores on the Asthma Control Questionnaire range from 0 to 6, with a higher score indicating worse asthma control.
Time Frame: The asthma control questionnaire score was measured on four occasions during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
units on a scale | -0.22 (0.055) | -0.31 (0.045) | -0.03 (0.048)

6. Secondary Outcome: Change Between Week 14 and Week 0 in the Albuterol Rescue Puffs Per Day
Description: Total number of puffs from the albuterol (rescue) inhaler during the previous 24 hours (excluding those puffs for preventive use).
Time Frame: Albuterol rescue puffs were measured daily during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: puffs per day
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
puffs per day | -0.11 (0.058) | -0.16 (0.063) | -0.07 (0.063)

7. Secondary Outcome: Change Between Week 14 and Week 0 in the Proportion of Asthma Control Days
Description: An asthma control day was defined as a day in which there were no symptoms and no albuterol (rescue) puffs.
Time Frame: An asthma control day was determined daily during each of the three 14-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: proportion of asthma control days
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Number analyzed (Participants) | 210 | 210 | 210
proportion of asthma control days | 0.13 (0.020) | 0.14 (0.023) | 0.05 (0.021)

ADVERSE EVENTS:
Time Frame: 1 year
Description: does not differ from clinicaltrials.gov definitions
Arm/Group | Tio + 1xICS | LABA + 1xICS | 2xICS
Serious Adverse Events (participants affected / at risk) | 3/203 | 4/196 | 4/195
Other Adverse Events (participants affected / at risk) | 2/203 | 2/196 | 6/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tio + 1xICS (N=203) | LABA + 1xICS (N=196) | 2xICS (N=195)
hospitalization due to pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
unrelated events (General disorders) | 1 (1) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tio + 1xICS (N=203) | LABA + 1xICS (N=196) | 2xICS (N=195)
urgent care visit due to asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
We evaluated only a small number of patients, with no treatment lasting longer than 14 weeks. We could not examine either the rate of asthma exacerbations or long-term safety issues, so our findings cannot be considered clinically directive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No